CLINICAL TRIAL: NCT01906879
Title: Comparison of the Efficacy of Clarithromycin-based Triple Therapy Versus Quadruple Therapies in the First Line Therapy of Helicobacter Pylori Infection- A Multicenter Randomized Comparative Trial
Brief Title: Triple Therapy Versus Quadruple Therapies in the First Line Therapy of Helicobacter Pylori Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201304017MINB
Record Dates: First submitted 2013-07-21; First posted 2013-07-24 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Triple therapy (A) (Active Comparator): lansoprazole, 30mg, twice daily, for 14 days, po clarithromycin, 500mg, twice daily, for 14 days, po amoxicillin, 1gm, twice daily, for 14 days, po
  Interventions: Drug: triple, quadruple, non-bismuth quadruple therapy
- non-bismuth quadruple therapy (Experimental): Group (B): non-bismuth quadruple therapy for 10 days: lansoprazole 30mg bid + amoxicillin 1gm bid + clarithromycin 500mg bid + metronidazole 500mg bid
  Interventions: Drug: triple, quadruple, non-bismuth quadruple therapy
- bismuth quadruple therapy for 10 days (Experimental): Group (C): bismuth quadruple therapy for 10 days D1-D10: lansoprazole 30mg bid + colloidal bismuth subcitrate 300mg tid + metronidazole 500mg tid + tetracycline 500mg tid
  Interventions: Drug: triple, quadruple, non-bismuth quadruple therapy

INTERVENTIONS:
Drug: triple, quadruple, non-bismuth quadruple therapy — triple therapy, quadruple therapy, non-bismuth quadruple therapy
  Other Names: Group (A): triple therapy for 14 days; Group (B): non-bismuth quadruple therapy for 10 days; Group (C): bismuth quadruple therapy for 10 days

SUMMARY:
Whether non-bismuth quadruple therapy (concomitant therapy) is more effective than bismuth quadruple therapy or triple therapy for 14 days remains unknown.

Therefore, we aim to compare the eradication rates and long term re-infection rates of quadruple therapy for 10 days versus non-bismuth quadruple therapy for 10 days vs. triple therapy for 14 days.

Methods: This will be a multi-center, open labeled, randomized control trial Patients: H. pylori infected patients who have willingness to receive eradication therapy

Testing for H. pylori infection Before First Line Ttreatment

(1)Any two positive of rapid urease test, histology, serology and culture or a positive UBT will be considered as H. pylori infected

After First Line Treatment: C13-Urea breath test will be used to assess the existence of H. pylori 6-8 weeks after first line therapy.

Long term reinfection: C13- Urea breath test will be used to assess the recurrence of H. pylori 1 year after eradication therapy

DETAILED DESCRIPTION:
First line therapy: open labeled, randomized control trial, randomized into one of the three groups Group (A): triple therapy for 14 days D1-D14: (lansoprazole 30mg + clarithromycin 500mg + amoxicillin 1gm) bid Group (B): non-bismuth quadruple therapy for 10 days D1-D10: lansoprazole 30mg bid + amoxicillin 1gm bid + clarithromycin 500mg bid + metronidazole 500mg bid Group (C): bismuth quadruple therapy for 10 days D1-D10: lansoprazole 30mg bid + colloidal bismuth subcitrate 300mg tid + metronidazole 500mg tid + tetracycline 500mg tid

Second line therapy: patients who fail from first line treatment will be rescue with the following treatment Group (A) Patient who fail from triple therapy will be retreated with bismuth quadruple therapy for 10 days D1-D10: lansoprazole 30mg bid + colloidal bismuth subcitrate 300mg tid + metronidazole 500mg tid + tetracycline 500mg tid Group (B) Patient who fail from non-bismuth quadruple therapy will be retreated with bismuth quadruple therapy for 10 days D1-D10: lansoprazole 30mg bid + colloidal bismuth subcitrate 300mg tid + metronidazole 500mg tid + tetracycline 500mg tid Group (C) Patients who fail from bismuth quadruple therapy will be retreated with non-bismuth quadruple therapy for 10 days D1-D10: lansoprazole 30mg bid + amoxicillin 1gm bid + clarithromycin 500mg bid + metronidazole 500mg bid

ELIGIBILITY:
Inclusion Criteria:

Patients aged greater than 20 years who have H. pylori infection without prior eradication therapy and are willing to receive the sequential therapy will be eligible for enrolment. Written informed consents will be obtained from all patients prior to enrollment.

Exclusion Criteria:

Patients will be excluded from the study if any one of the following criteria is present: (1) children and teenagers aged less than 20 years, (2) history of gastrectomy, (3)gastric malignancy, including adenocarcinoma and lymphoma, (4) previous allergic reaction to antibiotics (amoxicillin, clarithromycin, metronidazole, or levofloxacin) and prompt pump inhibitors (lansoprazole), (5)contraindication to treatment drugs, (6) pregnant or lactating women, (7) severe concurrent diseases, and (8) Patients who cannot give informed consent by himself or herself.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1620 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Eradication rate for H. pylori | 6 weeks
  Eradication rate in the first line according to intention to treat (ITT) and per-protocol (PP) analysis in the three treatment groups

SECONDARY OUTCOMES:
Adverse effects of each treatments | 2 weeks
  (1) Incidence of adverse effects in the first line therapy in the three treatment groups

OTHER OUTCOMES:
Reinfection rate | 1 year
  1. Eradication rates in the second line treatment in the three treatment groups
  2. Overall eradication rates after first line and second line treatment in the three treatment groups
  3. Antibiotic resistance of gut flora after first line and second line treatments in the three treatment groups
  4. Changes of gut microbiota in the three treatment groups
  5. Re-infection rate one year after eradication therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shiang Wu, MD. PhD, Principal Investigator — National Taiwan University Hospital, Taipei, Taiwan
Locations (10):
- Taiwan (10):
  - Chiayi Christian Hospital, Chiayi City
  - National Taiwan University Hospital, Hsinchu Branch, Hsinchu
  - E- DA Hospital and I-Shou University, Kaohsiung City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Ming-Shiang Wu, Taipei
  - Mackay Memorial Hospital, Taipei, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Mackay Memorial Hospital, Taitung, Taitung
  - National Taiwan University Hospital, Yun-Lin Branch, Yun-Lin County

REFERENCES:
- [Derived] Liou JM, Chen CC, Chang CM, Fang YJ, Bair MJ, Chen PY, Chang CY, Hsu YC, Chen MJ, Chen CC, Lee JY, Yang TH, Luo JC, Chen CY, Hsu WF, Chen YN, Wu JY, Lin JT, Lu TP, Chuang EY, El-Omar EM, Wu MS; Taiwan Gastrointestinal Disease and Helicobacter Consortium. Long-term changes of gut microbiota, antibiotic resistance, and metabolic parameters after Helicobacter pylori eradication: a multicentre, open-label, randomised trial. Lancet Infect Dis. 2019 Oct;19(10):1109-1120. doi: 10.1016/S1473-3099(19)30272-5. PMID 31559966
- [Derived] Liou JM, Fang YJ, Chen CC, Bair MJ, Chang CY, Lee YC, Chen MJ, Chen CC, Tseng CH, Hsu YC, Lee JY, Yang TH, Luo JC, Chang CC, Chen CY, Chen PY, Shun CT, Hsu WF, Hu WH, Chen YN, Sheu BS, Lin JT, Wu JY, El-Omar EM, Wu MS; Taiwan Gastrointestinal Disease and Helicobacter Consortium. Concomitant, bismuth quadruple, and 14-day triple therapy in the first-line treatment of Helicobacter pylori: a multicentre, open-label, randomised trial. Lancet. 2016 Nov 12;388(10058):2355-2365. doi: 10.1016/S0140-6736(16)31409-X. Epub 2016 Oct 18. PMID 27769562